CLINICAL TRIAL: NCT07363031
Title: Characterization of the Herpesviridae Family in the Oral Cavity and Its Association With Oral Mucositis in Adult Patients Undergoing Head and Neck Radiotherapy: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Prophylactic Valacyclovir
Brief Title: Oral Herpesviruses and Oral Mucositis in Patients Receiving Head and Neck Radiotherapy
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Oncoclinicas (Other)
Collaborators: Oswaldo Cruz Foundation (Other); Hospital Sírio-Libânes, São Paulo, Brazil (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 56941822.3.0000.5134
Record Dates: First submitted 2026-01-08; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Oral Mucositis; Head and Neck Cancer (H&N); Radiotherapy Side Effects
Keywords: Oral Mucositis; Head and Neck Cancer; Radiotherapy; Herpesviridae; Herpesvirus reactivation; Valacyclovir; Antiviral prophylaxis; Oral toxicity; Supportive care in oncology; Randomized controlled trial
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms | interventions — Valacyclovir

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups to receive either prophylactic valacyclovir or placebo during radiotherapy for head and neck cancer. Each participant remains in the assigned group for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, healthcare providers, investigators, and outcome assessors are blinded to treatment allocation. Valacyclovir and placebo are identical in appearance and administration, and treatment assignment is concealed until completion of data analysis or in the event of a medical emergency requiring unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Valacyclovir (Experimental): Participants in this arm receive oral valacyclovir during radiotherapy for head and neck cancer to evaluate its effect on oral herpesvirus detection and oral mucositis outcomes.
  Interventions: Drug: Valacyclovir
- Placebo (Placebo Comparator): Participants in this arm receive a matching placebo during radiotherapy for head and neck cancer for comparison with the valacyclovir group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir — Valacyclovir is administered orally during the course of radiotherapy for head and neck cancer as a prophylactic antiviral intervention.
  Arms: Valacyclovir
Drug: Placebo — A matching placebo is administered orally during the course of radiotherapy for head and neck cancer.
  Arms: Placebo

SUMMARY:
Patients receiving radiotherapy for head and neck cancer often develop oral mucositis, a painful condition that causes redness and sores in the mouth. Oral mucositis can make it difficult to eat, drink, and speak, and may interfere with cancer treatment. Some viruses from the herpesvirus family, which commonly remain inactive in the body, may become active during cancer treatment and worsen mouth sores. However, the role of these viruses in oral mucositis is not fully understood.

This study aims to understand whether herpesviruses present in the mouth are associated with the development and severity of oral mucositis in adults receiving radiotherapy for head and neck cancer. The study also evaluates whether taking an antiviral medication (valacyclovir) can reduce viral activity and improve mouth symptoms during treatment.

Participants are randomly assigned to receive either valacyclovir or a placebo while undergoing radiotherapy. Samples from the mouth and saliva are collected at different time points before, during, and after radiotherapy to detect herpesviruses. Mouth sores are regularly examined, and pain levels are recorded throughout treatment.

The results of this study may help clarify the role of herpesviruses in oral mucositis and support better strategies to prevent or manage this condition in patients receiving radiotherapy for head and neck cancer.

DETAILED DESCRIPTION:
Oral mucositis is a frequent and clinically significant side effect of radiotherapy for head and neck cancer. While mucosal injury is primarily related to radiation exposure, additional biological factors may influence the onset and severity of this condition. Reactivation of viruses from the Herpesviridae family has been suggested as a potential contributing factor, but existing evidence is limited and inconsistent. There is currently no standard preventive antiviral strategy for oral mucositis in this population.

This study is designed to characterize the presence and changes of herpesviruses in the oral cavity of adults undergoing radiotherapy for head and neck cancer and to evaluate whether prophylactic antiviral treatment affects viral detection and clinical outcomes related to oral mucositis. The trial uses a randomized, double-blind, placebo-controlled design to reduce bias and allow for an objective assessment of antiviral prophylaxis.

Participants receive either oral valacyclovir or matching placebo during the course of radiotherapy. Oral and saliva samples are collected at predefined time points before the start of radiotherapy, during treatment, and after completion of radiotherapy. These samples are analyzed to detect and quantify human herpesviruses using molecular methods. Clinical assessments of the oral cavity are performed regularly to evaluate the presence and severity of oral mucositis, and patient-reported pain is monitored throughout treatment.

The study aims to describe the pattern of herpesvirus detection in the oral cavity over time and to explore associations between viral presence, mucositis severity, and pain. In addition, the study evaluates whether antiviral prophylaxis influences these outcomes when compared with placebo.

By improving the understanding of the relationship between herpesvirus activity and oral mucositis, this study may inform future preventive or supportive care strategies for patients receiving radiotherapy for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosis of head and neck cancer.
* Planned to receive curative or definitive radiotherapy to the head and neck region.
* Ability to swallow oral medication.
* Adequate clinical condition to participate in study procedures.
* Ability to provide written informed consent.

Exclusion Criteria:

* Known hypersensitivity or contraindication to valacyclovir or related antiviral agents.
* Current or recent use of systemic antiviral therapy.
* Severe renal impairment requiring dose adjustment or contraindicating valacyclovir use.
* Active oral infection requiring systemic antimicrobial treatment at baseline.
* Pregnant or breastfeeding individuals.
* Participation in another interventional clinical trial that may interfere with study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Severity of Oral Mucositis | From start of radiotherapy (day 1) until 2 weeks after completion of radiotherapy.
  Maximum oral mucositis severity assessed using the World Health Organization (WHO) Oral Mucositis Grading Scale, which ranges from 0 (no mucositis) to 4 (severe mucositis). Higher scores indicate worse oral mucositis severity.

SECONDARY OUTCOMES:
Incidence of Ulcerative Oral Mucositis | From start of radiotherapy (Day 1) until 2 weeks after completion of radiotherapy.
  Proportion of participants who develop ulcerative oral mucositis (World Health Organization [WHO] Oral Mucositis Grading Scale grade ≥ 2) during radiotherapy. The WHO Oral Mucositis Grading Scale ranges from 0 (no mucositis) to 4 (severe mucositis), with higher scores indicating worse oral mucositis severity.

OTHER OUTCOMES:
Oral Pain Intensity | From start of radiotherapy (Day 1) until 2 weeks after completion of radiotherapy.
  Oral pain intensity measured using the Numeric Rating Scale for Pain, ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicate worse pain intensity.
Oral Herpesvirus Detection and Viral Load Over Time | From start of radiotherapy (Day 1), weekly during radiotherapy, and 1 month after completion of radiotherapy (approximately up to 12 weeks).
  Presence and quantitative viral load of human herpesviruses in oral and saliva samples measured using real-time polymerase chain reaction (qPCR).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Oncoclinicas, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results of this study will be made available upon reasonable request. Requests will be reviewed by the study investigators and subject to institutional approvals and data sharing agreements, in accordance with ethical and regulatory requirements.
Supporting Information: Study Protocol
Time Frame: De-identified individual participant data and the study protocol will be available beginning after publication of the primary study results and will remain available for up to 5 years following publication.
Access Criteria: Access to de-identified individual participant data and the study protocol will be provided to qualified researchers upon reasonable request. Requests will be reviewed by the study investigators and subject to approval by the sponsoring institution, execution of a data use agreement, and compliance with ethical and regulatory requirements. Only data necessary to achieve the approved research objectives will be shared.